CLINICAL TRIAL: NCT00444184
Title: A Crossover, Double-Masked Comparison Investigating the 24-Hour Intraocular Pressure Control With the Travoprost/Timolol Fixed Combination Versus Travoprost, When Both Are Given in the Evening, in Subjects With Primary Open-Angle Glaucoma
Brief Title: 24-hour Intraocular Pressure Control With Travoprost/Timolol Fixed Combination Versus Travoprost
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A3243
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma
Keywords: travoprost/timolol fixed combination
MeSH Terms: conditions — Glaucoma | interventions — Travoprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost/Timolol therapy (Active Comparator): 24-hour pressure monitoring after 3 months of chronic dosing with travoprost/timolol drops
  Interventions: Drug: Travoprost/timolol fixed combination, travoprost
- Travoprost therapy (Active Comparator): 24-hour pressure monitoring after 3 months of chronic dosing with travoprost drops
  Interventions: Drug: Travoprost/timolol fixed combination, travoprost

INTERVENTIONS:
Drug: Travoprost/timolol fixed combination, travoprost

SUMMARY:
This 8-week, crossover study will compare the quality of 24-hour IOP control with TTFC versus travoprost when both medications are dosed in the evening. Such a crossover comparison may determine the real efficacy of the new fixed combination versus travoprost monotherapy. The results should enhance the investigators understanding on the best dosing of TTFC and may influence its clinical use in Europe. Finally, the results would better delineate the future role of TTFC in glaucoma management after PG monotherapy, or instead of unfixed therapy with PG analogs and timolol. This study should assist the general ophthalmologist worldwide to plan optimal stepwise medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adults with primary open-angle glaucoma (POAG) who exhibit a mean untreated IOP greater than 23 m Hg at baseline (10:00).
* Patient has POAG and is older than 29 years
* The IOP without treatment is greater than 23 mm Hg and lower than 38 mm Hg at baseline (2 readings at 10:00)
* Patient can be safely washed out without risk for significant deterioration
* Distance best corrected Snellen visual acuity better than 1/10
* Patient can understand the instructions and comply to medications
* Open normal appearing angles

Exclusion Criteria:

* Contraindications to prostaglandins or β-blockers
* History of lack of response (<10% reduction) to any medication
* Female of childbearing potential or lactating mother
* History of trauma, inflammation, surgery, past use of steroids (within 2 months), severe dry eyes and use of contact lenses
* Sign of ocular infection, except blepharitis, corneal abnormality that may affect IOP measurements etc

Ages: 29 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Mean 24-hour IOP | 3 months

SECONDARY OUTCOMES:
Mean reduction from baseline | 3 months
Mean fluctuation of 24-hour IOP | 3 months
Individual IOP readings measured at 10:00 (± 1 hour) and at +4, +8, +12, +16 and +20 (± 1 hour) hours. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios GP Konstas, MD, PhD, Principal Investigator — Associate Professor and Head of the Glaucoma Unit, 1st University Department of Ophthalmology
Locations (1):
- Glaucoma Unit, 1st University Department of Ophthalmology, Thessaloniki, Greece